CLINICAL TRIAL: NCT06908577
Title: A Multiple Centre, Randomised, Open-label, Parallel Group, Phase I Pharmacokinetic Comparability Study of Tozorakimab Administered Using an Accessorised Prefilled Syringe (APFS) or an Autoinjector (AI) in Healthy Volunteers
Brief Title: An Accessorised Prefilled Syringe to an Autoinjector Pharmacokinetic Bridging Study of Tozorakimab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9180C00006; 2024-511840-22 (Other: EU CT Number); 2024-511840-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-04-02; First posted 2025-04-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Anti-Interleukin (IL)-33 antibody; Human immunoglobulin G1 monoclonal antibody; Accessorised Prefilled Syringe (APFS); Autoinjector (AI); Respiratory and Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Tozorakimab (Test) (Experimental): Participants will receive a single SC dose of tozorakimab via AI device.
  Interventions: Drug: Tozorakimab; Device: Autoinjector (AI) Device
- Treatment B: Tozorakimab (Reference) (Active Comparator): Participants will receive a single SC dose of tozorakimab via APFS device with the same container closure as the AI.
  Interventions: Drug: Tozorakimab; Device: Accessorised Prefilled Syringe (APFS) Device

INTERVENTIONS:
Drug: Tozorakimab — Tozorakimab will be administered as a single SC dose using an AI or APFS device on Day 1.
  Other Names: MEDI3506
Device: Autoinjector (AI) Device — AI device will be used to administer single SC dose of tozorakimab on Day 1.
  Arms: Treatment A: Tozorakimab (Test)
Device: Accessorised Prefilled Syringe (APFS) Device — APFS device will be used to administer single SC dose of tozorakimab on Day 1.
  Arms: Treatment B: Tozorakimab (Reference)

SUMMARY:
The purpose of this study is to compare the pharmacokinetic (PK) exposures of a single subcutaneous (SC) dose of tozorakimab administered using AI or APFS in healthy participants.

DETAILED DESCRIPTION:
This is a multiple center, randomized, open-label, parallel group, Phase 1 study.

Participants will be randomized 1:1:1:1:1:1 to one of the 6 combinations of the devices (APFS or AI devices) and one of three injection sites (abdomen, thigh, or upper arm.).

The study includes:

* A screening period of up to 28 days.
* A treatment period (up to 9 days).
* A follow-up period till 85 days.
* A final follow-up visit on Day 113 (Week 16).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the screening visit and on admission.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception, in order to avoid pregnancy from the time of administration of study intervention until 16 weeks after administration of the study intervention (Day 113).
* Females of non-childbearing potential must be confirmed at the screening visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods from the time of administration of the study intervention until 16 weeks after administration of the study intervention (Day 113).
* Have a body mass index (BMI) between 19 and 30 kg/m2 inclusive and weigh at least 55 kg and no more than 100 kg inclusive at screening and Day -1.
* Intact normal skin without potentially obscuring tattoos, scars, etc., at the injection site.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results of the study or the participant's ability to participate in the study.
* Any clinically important medical/surgical procedure or trauma within 8 weeks of the screening visit, or any planned inpatient hospitalization during the study period.
* Malignancy, current or within the past 5 years, suspected malignancy or undefined neoplasms.
* Any abnormal laboratory values and vital signs.
* History of known immunodeficiency disorder, including a positive test for human immunodeficiency virus (HIV)-1 or HIV-2.
* History or treatment for hepatitis B or hepatitis C or any positive test result on screening for hepatitis B surface antigen (HBsAg), anti-hepatitis B core (HBc) antibodies, or anti-hepatitis C antibodies.
* Evidence of currently active tuberculosis (TB) disease or use of any TB drug treatment in the past 12 months or latent TB infection.
* Any clinically significant abnormalities on 12lead electrocardiogram (ECG) at the screening visit and/or admission (Day -1) to the Clinical Unit.
* History of or ongoing severe clinically important allergy/hypersensitivity, or history of hypersensitivity to monoclonal or polyclonal antibodies. History of allergy or reaction to any formulation components of the investigational medicinal product (IMP).
* Receipt of live attenuated vaccines within 30 days prior to randomization and receipt of COVID-19 or inactivated vaccines within 14 days prior to randomization.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months or 5 half-lives of time of dosing in this study, whichever is longer.
* Receipt of any investigational biologic within 4 months or 5 half-lives prior to the date of dosing in this study, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) of tozorakimab | From Day 1 to Day 113
  To compare the PK exposure following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of tozorakimab | From Day 1 to Day 113
  To compare the PK exposure following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Maximum observed drug concentration (Cmax) of tozorakimab | From Day 1 to Day 113
  To compare the PK exposure following single SC administration of tozorakimab using AI and APFS devices in healthy participants.

SECONDARY OUTCOMES:
Time to reach maximum observed concentration (Tmax) | From Day 1 to Day 113
  To assess additional PK parameters following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Terminal elimination half-life (t1/2λz) | From Day 1 to Day 113
  To assess additional PK parameters following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Terminal rate constant (λz) | From Day 1 to Day 113
  To assess additional PK parameters following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Apparent total body clearance (CL/F) | From Day 1 to Day 113
  To assess additional PK parameters following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Apparent volume of distribution based on the terminal phase (Vz/F) | From Day 1 to Day 113
  To assess additional PK parameters following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Number of participants with adverse events (AEs) | From screening (Day -28 to -2) to follow up (Day 113)
  To assess the safety and tolerability following single SC administration of tozorakimab using AI and APFS devices in healthy participants.
Number of participants with positive anti-drug antibodies (ADA) | From Day 1 to Day 113
  To evaluate the immunogenicity following single SC administration of tozorakimab using AI and APFS devices in healthy participants.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland
- Research Site, Berlin, Germany
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/